CLINICAL TRIAL: NCT05839834
Title: A Blinded Prospective Study on Development and Validation of the Blood Cell RNA-Based Cancer Detection
Brief Title: Blood Cell RNA-Based Cancer Detection
Acronym: eRBCDet
Status: Recruiting | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Zheng Wang, MD/PhD, Study chair, Clinical Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: blood-cell-RNA
Record Dates: First submitted 2022-07-12; First posted 2023-05-03 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Neoplasms; Cancer
MeSH Terms: conditions — Neoplasms | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer: Patients with new diagnosis of cancers
  Interventions: Diagnostic Test: Blood test
- Non-cancer: Healthy participants
  Interventions: Diagnostic Test: Blood test

INTERVENTIONS:
Diagnostic Test: Blood test — RNA sequencing of peripheral blood cells

SUMMARY:
Early diagnosis of cancer may provide patients with more treatment options and hopefully prolong survival. The purpose of this multi-center study is to collect peripheral blood from newly diagnosed cancer patients and healthy donors to establish a blood cell RNA-based model for the differentiation of cancer patients and healthy donors. The area under the receiver operating characteristic (AUROC), sensitivity and specificity of the test in the early detection of multiple cancers will be measured.

ELIGIBILITY:
Inclusion Criteria for All the Participants

1. Age 18 years or older
2. Provide informed consent

Exclusion Criteria for All the Participants:

1. Pregnancy or lactating women
2. Received a blood transfusion within 1 month
3. Received anti-cancer treatment within 3 years
4. Known prior diagnosis of cancer
5. Poor health status or unfit to tolerate blood draw

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed cancer patients and healthy donors will be recruited from medical centers.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-02-08 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-08 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of cancer detection | 1 year
  Sensitivity and specificity of the early detection of 30 types of cancers of a blood cell RNA-based cancer detection test
Accuracy of TOO prediction | 1 year
  Accuracy of the tissue of origin (TOO) prediction of a blood cell RNA-based cancer detection test

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Wang, MD/PhD, Study Chair — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Zheng Wang, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mellby LD, Nyberg AP, Johansen JS, Wingren C, Nordestgaard BG, Bojesen SE, Mitchell BL, Sheppard BC, Sears RC, Borrebaeck CAK. Serum Biomarker Signature-Based Liquid Biopsy for Diagnosis of Early-Stage Pancreatic Cancer. J Clin Oncol. 2018 Oct 1;36(28):2887-2894. doi: 10.1200/JCO.2017.77.6658. Epub 2018 Aug 14. PMID 30106639
- [Background] Liu MC, Oxnard GR, Klein EA, Swanton C, Seiden MV; CCGA Consortium. Sensitive and specific multi-cancer detection and localization using methylation signatures in cell-free DNA. Ann Oncol. 2020 Jun;31(6):745-759. doi: 10.1016/j.annonc.2020.02.011. Epub 2020 Mar 30. PMID 33506766
- [Background] Klein EA, Richards D, Cohn A, Tummala M, Lapham R, Cosgrove D, Chung G, Clement J, Gao J, Hunkapiller N, Jamshidi A, Kurtzman KN, Seiden MV, Swanton C, Liu MC. Clinical validation of a targeted methylation-based multi-cancer early detection test using an independent validation set. Ann Oncol. 2021 Sep;32(9):1167-1177. doi: 10.1016/j.annonc.2021.05.806. Epub 2021 Jun 24. PMID 34176681
- [Background] Best MG, Sol N, In 't Veld SGJG, Vancura A, Muller M, Niemeijer AN, Fejes AV, Tjon Kon Fat LA, Huis In 't Veld AE, Leurs C, Le Large TY, Meijer LL, Kooi IE, Rustenburg F, Schellen P, Verschueren H, Post E, Wedekind LE, Bracht J, Esenkbrink M, Wils L, Favaro F, Schoonhoven JD, Tannous J, Meijers-Heijboer H, Kazemier G, Giovannetti E, Reijneveld JC, Idema S, Killestein J, Heger M, de Jager SC, Urbanus RT, Hoefer IE, Pasterkamp G, Mannhalter C, Gomez-Arroyo J, Bogaard HJ, Noske DP, Vandertop WP, van den Broek D, Ylstra B, Nilsson RJA, Wesseling P, Karachaliou N, Rosell R, Lee-Lewandrowski E, Lewandrowski KB, Tannous BA, de Langen AJ, Smit EF, van den Heuvel MM, Wurdinger T. Swarm Intelligence-Enhanced Detection of Non-Small-Cell Lung Cancer Using Tumor-Educated Platelets. Cancer Cell. 2017 Aug 14;32(2):238-252.e9. doi: 10.1016/j.ccell.2017.07.004. PMID 28810146
- [Background] Best MG, Sol N, Kooi I, Tannous J, Westerman BA, Rustenburg F, Schellen P, Verschueren H, Post E, Koster J, Ylstra B, Ameziane N, Dorsman J, Smit EF, Verheul HM, Noske DP, Reijneveld JC, Nilsson RJA, Tannous BA, Wesseling P, Wurdinger T. RNA-Seq of Tumor-Educated Platelets Enables Blood-Based Pan-Cancer, Multiclass, and Molecular Pathway Cancer Diagnostics. Cancer Cell. 2015 Nov 9;28(5):666-676. doi: 10.1016/j.ccell.2015.09.018. Epub 2015 Oct 29. PMID 26525104